CLINICAL TRIAL: NCT06020716
Title: A Phase 4 Double Blinded Study With Two Different Interventions, Each With Two Arms, to Evaluate the Clinical Efficacy of Antibiotics and the Role of Microbiology, Immunology and Genetics in Children Aged 9-36 Months With Chronic Wet Cough.
Brief Title: Antibiotics, Microbiology and Immunology in Children With Chronic Wet Cough - the AMIC Study
Acronym: AMIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Oslo University Hospital (Other); Haukeland University Hospital (Other); Alesund Hospital (Other); University Hospital, Akershus (Other); Trondheim University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMIC 2023; 2022-500586-27-00 (Other: EU CT number)
Record Dates: First submitted 2023-07-03; First posted 2023-09-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Protracted Bacterial Bronchitis
Keywords: Chronic wet cough; Antibiotic; Children; Microbiology; Immunology
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: This is a Phase 4, randomized controlled, parallel group, multicenter, double blind study of amoxicillin-clavulanate in children 9-36 months of age with chronic wet cough. A total of 300 children will be included in the study in two different RCTs; AMIC 1 and AMIC 2.AMIC 1 will be performed before AMIC 2.There is no randomization between AMIC 1 and AMIC 2.
  To study the role of respiratory pathogens, microbiome and inflammation, 50 healthy controls will be included for comparison.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AMIC 1: Arm A (Experimental): In AMIC 1, 90 children will be randomly be assigned 1:1 to receive either amoxicillin-clavulanate syrup or placebo (Arm A and B) for 14 days. AMIC 1 Arm A will receive 14 days amoxicillin-clavulanate syrup.
  Interventions: Drug: Amoxicillin-Clavulanate 400 Mg-57 Mg/5 mL Oral Powder for Reconstitution
- AMIC 1: Arm B (Placebo Comparator): In AMIC 1, 90 children will be randomly be assigned 1:1 to receive either amoxicillin-clavulanate syrup or placebo (arm A and B) for 14 days. AMIC 1 Arm B will receive 14 days placebo syrup.
  Interventions: Drug: Placebo
- AMIC 2: Arm C (Experimental): In AMIC 2, 210 children will be randomly assigned 1:1 to receive either 14 or 28 days with amoxicillin-clavulanate syrup (arm C and D). AMIC 2 Arm C will receive 14 days amoxicillin-clavulanate syrup and 14 days placebo.
  Interventions: Drug: Amoxicillin-Clavulanate 400 Mg-57 Mg/5 mL Oral Powder for Reconstitution; Drug: Placebo
- AMIC 2: Arm D (Experimental): In AMIC 2, 210 children will be randomly assigned 1:1 to receive either 14 or 28 days with amoxicillin-clavulanate syrup (arm C and D). AMIC 2 Arm D will receive 28 days amoxicillin-clavulanate syrup.
  Interventions: Drug: Amoxicillin-Clavulanate 400 Mg-57 Mg/5 mL Oral Powder for Reconstitution

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate 400 Mg-57 Mg/5 mL Oral Powder for Reconstitution — Three times daily
  Arms: AMIC 1: Arm A; AMIC 2: Arm C; AMIC 2: Arm D
Drug: Placebo — Three times daily
  Arms: AMIC 1: Arm B; AMIC 2: Arm C

SUMMARY:
The AMIC study is a double-blind, placebo-controlled, multicenter, nationwide, randomized controlled academic pharmaceutical trial.

OVERALL PRIMARY OBJECTIVES:

* To study the clinical efficacy of antibiotics in children with chronic wet cough (CWC).
* To study if duration of treatment with antibiotics in children with CWC has impact on efficacy or time to relapse of symptoms.

OVERALL SECONDARY OBJECTIVE:

-To study respiratory pathogens and the diversity/composition of airway and gut microbiome in children with CWC compared to healthy controls, and changes in pathogens/microbiome after treatment with antibiotics.

OVERALL TERTIARY OBJECTIVE:

-To study the role of inflammation, immunology, and genetics in children with chronic wet cough and suspicion of PBB to increase the knowledge of pathophysiological mechanisms associated with PBB.

The study will include two different RCTs AMIC 1 and AMIC 2:

AMIC 1:

Participants will be randomly assigned to 14 days amoxicillin-clavulanate syrup or placebo.

AMIC 2:

Participants will be randomly assigned 1:1 to receive either 14 or 28 days with amoxicillin-clavulanate syrup.

DETAILED DESCRIPTION:
Study populations:

AMIC 1:

90 children with chronic wet cough aged 9-36 months.

AMIC 2:

210 children with chronic wet cough aged 9-36 months.

All children will be followed until 24 months after the start of the Randomized Controlled Trial (RCT).

HEALTHY CONTROL GROUP:

To study the role of respiratory pathogens, airway and gut microbiome, inflammation and immunology, 50 healthy controls will be included for comparison to AMIC 1. The healthy controls will have a second visit 6 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 9 and < 36 months.
2. Body weight ≥ 7 kg and < 24 kg.
3. Born term with Gestational age ≥ 37 weeks.
4. Chronic wet cough for > 4 weeks at screening and in addition average cough score last 7 days at randomization ≥ 4 points and without signs of another cause. Registration ≥ 5 days is mandatory.
5. Written informed consent obtained from both parents at inclusion.
6. The study subject must be assessed as eligible for treatment with Augmentin.

Exclusion Criteria:

1. Gestational age < 37 weeks.
2. History of acute upper or lower airway infection the last 2 weeks.
3. History of other viral or bacterial infections the last 2 weeks.
4. Episode with temperature above 38 °C during the last 2 weeks.
5. Previous diagnosed with chronic lung disease such as cystic fibrosis, primary ciliary dyskinesia, interstitial lung disease, asthma, immunodeficiency, esophagus atresia.
6. Cardiac disease, except persisting foramen ovale or ductus arteriosus.
7. Severe feeding problems/aspiration.
8. Gastroesophageal reflux suspicion or confirmed by ph measurement.
9. Suspicion of hypertrophic tonsils or adenoids
10. Episodes of bronchopulmonary obstruction suggesting asthma
11. Presence of gross neurodevelopmental delay, or suspicion of neurological disease.
12. History of known or suspected allergic reactions to amoxicillin-clavulanate or any other betalactam.
13. Episodes with haemoptysis and with unknown cause.
14. Radiographic changes other than perihilar changes confirmed by x-ray at screening.
15. At examination: Digital clubbing, hypoxia, chest wall deformity, dyspnoea at rest.
16. Parents unable to speak and/or understand Norwegian language.
17. Received systemic antibiotics within the last 6 months before inclusion.
18. Participation in another clinical intervention trial.

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | Response to treatment will be assessed 14 days after end of antibiotic treatment
  Response to treatment is defined as an improvement in baseline validated Verbal category descriptive (VCD) cough score ≤2 at the end of treatment or cessation of coughing for a minimum period of 3 days within the treatment period.The VCD score has a minimum and maxiumum score ranging from 0-10 points, and a higher value corresponds to more severe cough.

SECONDARY OUTCOMES:
Relapse of symptoms | Relapse of symptoms will be assessed up to 24 months after end of antibiotic treatment
  Relapse of symptoms after antibiotic treatment for chronic wet cough is defined as a new period of wet cough - after a period of at least 7 days without symptoms - lasting for more than four weeks, or an episode of wet cough of at least two weeks duration which was treated with antibiotics by the child's general practitioner or treating physician. The start of relapse is the first day of cough of such a period or episode.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Øymar, MD PhD, Study Chair — Helse Stavanger HF
Locations (7):
- Norway (7):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lillestrøm
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North-Norway, Tromsø
  - Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No